CLINICAL TRIAL: NCT02898831
Title: Cold Compress for Pain Associated With Intrauterine Device Insertion: A Randomized Controlled Trial
Brief Title: Cold Compress for Pain Associated With Intrauterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20004308
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2018-01

CONDITIONS: Intrauterine Device; Cold Compress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control/No Intervention (No Intervention): Standard clinical procedure with intrauterine device insertion involving no heated/cold compresses on the abdomen during insertion.
- Cold Compress/Experimental (Experimental): Cold compress (intervention) placed on abdomen just before IUD insertion and remains throughout insertion. Pain scale and survey completed following insertion regarding pre-procedure and intra-procedure pain.
  Interventions: Other: Cold Compress

INTERVENTIONS:
Other: Cold Compress — Cold Compress placed on lower abdomen prior to and during IUD insertion.
  Other Names: Ice Pack
  Arms: Cold Compress/Experimental

SUMMARY:
This study will be a prospective randomized controlled trial comparing cold compression to no intervention immediately prior to and during intrauterine device insertion. Subjects will be randomized to cold compress or no intervention (standard practice in our clinics). Following IUD insertion they will complete a validated pain scale survey regarding their pre-procedure and intra-procedure pain.

DETAILED DESCRIPTION:
This study will be a prospective randomized controlled trial comparing cold compression to no intervention immediately prior to and during intrauterine device insertion. Inclusion criteria include all non-pregnant women, 18 years of age or older, presenting to the VCU Women's Health clinics with desired IUD placement.

Subjects will be identified at the time of presentation to the Women's Health Clinics at Virginia Commonwealth University Health Systems. A provider (physician, nurse practioner, or nurse midwife) will discuss the study with the subject. After time for consideration and having had all questions answered the subject will then be consented for the trial. Consent will be obtained at that time (see attached list of engaged providers). Randomization will be performed by pulling sequentially numbered opaque envelopes containing computer randomized individual allocations. This randomization will be carried out by research staff before the initiation of the study. Information regarding basic demographic data, comorbidities that may affect patient's perception of pain will be obtained from the subjects' chart. This information will include: age, race, socioeconomic status, status of practitioner, parity, BMI, history of prior cervical procedures, history of chronic pain.

If the subject has elected to participate in study and is randomized to the cold compression group, she will have a cold compress placed on the abdomen five minutes prior to and throughout the intrauterine device placement. Visual acuity pain scales have been commonly used in similar studies to objectively assess procedural pain. In this study, a validated 10 point visual acuity scale will be used. Pain will be assessed pre- and post-procedure. The post-procedure questions are directed at pain during the procedure.

Comparable studies that assess procedural pain considered a 30% reduction in pain to be significant. Based on these studies we will similarly consider a 30% reduction in pain between the experimental and control groups to be significant. With a power of 80 and significance value of p < 0.05, this will require 69 patients in each group (cold compression versus no-intervention) to obtain an adequate sample size to detect a difference in the groups. The study was powered for the post-treatment means of the control groups to be 2.8 and 4.0 (respectively), which is a 30% difference, assuming a SD=2.8 and using a two-sample t-test. Paper copies of written consent and any identifying information will be kept in a secured, locked file. All data collected will be stored in a password protected computer file that will be accessible only to the investigators.

The primary outcome will be the difference in patient's perception of pain before and during intrauterine device insertion. This will be defined based on a pre and post-procedure survey using a 10-point visual analogue scale. Additionally, nulliparous and multiparous women will be stratified as previous studies have shown significantly different pain scores reported between these two subgroups.

The investigators will collect the data, perform data entry and review charts to ensure accuracy of information provided by the inserting physician. Periodic review of the data entry will be performed to ensure completeness and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant women,
* 18 years of age or older,
* desire IUD placement.

Exclusion Criteria:

* under the age of 18
* decisionally impaired
* prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Procedural Pain | During IUD insertion (second to minutes)
  Primary outcome will be the difference in patient's perception of pain before and during intrauterine device insertion. This will be defined based on a pre and post-procedure survey using a 10-point visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - VCU Health System- Stony Point Clinic, Richmond, Virginia
  - VCU Health System Nelson Clinic, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Plan to make data visable on clinicaltrials.gov at the conclusion of the study.